CLINICAL TRIAL: NCT02607826
Title: Short-term Starvation vs. Normal Diet Before Chemotherapy of Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Michael Hötker, Dr. med., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Starvation Study
Record Dates: First submitted 2015-11-04; First posted 2015-11-18 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Cholangiocarcinoma; Pancreatic Ductal Adenocarcinoma; Colorectal Cancer; Gastric Cancer; Adenocarcinoma of the Esophagogastreal Junction; Esophagus Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Procedure: Starvation
- Standard of Care (No Intervention)

INTERVENTIONS:
Procedure: Starvation — Short-term starvation for a timeframe beginning 24h prior to chemotherapy administration, lasting until 6h after administration
  Arms: Intervention arm

SUMMARY:
Recent pre-clinical data provide strong evidence that short-term starvation before the administration of cytostatic drugs for the chemotherapy of solid tumors leads to significantly higher efficacy and lower toxicity levels. However, these findings have so far not been validated in patients. The aim of this trial is to provide first clinical evidence regarding the impact of pre-chemotherapeutic short-term starvation on response to therapy (primary endpoint). Additionally, progression-free survival, adverse events, and overall survival will be monitored (secondary endpoints). In perspective, short-term starvation before chemotherapy could represent a simple and secure way to improve both efficacy and tolerance of chemotherapies at low cost.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (male/female) ≥ 18 years of age
2. Written informed consent obtained prior to any trial specific procedure
3. Patient suffering from gastrointestinal tumors: Cholangiocarcinoma (CC), Pancreatic ductal adenocarcinoma (PDAC), Colorectal Cancer (CRC), Gastric Cancer (GC)/ Adenocarcinoma of the Esophagogastreal Junction (AEG) / Esophagus cancer (EC).
4. Planned to receive palliative chemotherapy
5. No prior palliative chemotherapy
6. ECOG performance status of 0 or 1
7. Life expectancy of 12 weeks or more
8. Adequate hematological parameters, as demonstrated by:

   * Hemoglobin > 9.0 g/dl (5.6 mmol/l)
   * WBC ≥ 3.0 x 109/l
   * ANC ≥ 1500/mm³
   * Platelets ≥ 75 x 109/l
   * S-creatinine ≤ 1.5 mg/dl (132 µmol/l)

Exclusion Criteria:

1. Underweight (BMI < 18.5)
2. Dysphagia
3. Insulin-dependent diabetes mellitus
4. Renal failure requiring hemo- or peritoneal dialysis
5. Pregnant or breast-feeding women
6. Drug/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Response to therapy on MRI or CT scancs will be measured using the RECIST criteria version 1.1. | Three Months
  Primary endpoint of this study is to assess the improvement in response to therapy for patients undergoing short-term starvation before chemotherapy of solid tumors in comparison to patients without dietary restrictions. Response to therapy on MRI or CT scancs will be measured using the RECIST criteria version 1.1.